CLINICAL TRIAL: NCT06983392
Title: Levels and Persistence of Oral DNA Adducts in Smokers, Vapers, and Non-users
Brief Title: Persistence of Oral DNA Adducts in Smokers and Vapers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025LS003
Record Dates: First submitted 2025-04-14; First posted 2025-05-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Smokers; Vaping; Healthy Volunteers
Keywords: smoking; vaping; tobacco; nicotine; abstain
MeSH Terms: conditions — Vaping; Smoking | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Participants will be asked to fill out study questionnaires and attend six in-person study visits to provide saliva, mouth cells, cheek cells, and urine. They will not be able to eat or drink anything other than water for at least 1 hour before your study visits.
  They may be asked to stop smoking cigarettes or vaping during the study for 21 days. If they are asked to abstain from their product use they will be given nicotine patches and/or lozenges to help with abstinence during the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Abstain from product use (either smoking cigarettes or vaping)
  Interventions: Behavioral: Abstain from smoking/vaping

INTERVENTIONS:
Behavioral: Abstain from smoking/vaping — They may be asked to stop smoking cigarettes or vaping during the study for 21 days. If they are asked to abstain from their product use they will be given nicotine patches and/or lozenges to help with abstinence during the study.

SUMMARY:
This study aims to better understand what damage caused to oral cells from smoking and vaping might be important in the formation of oral cancers. We will compare levels of DNA damage between those asked to stop smoking or vaping to those who continue to smoke or vape and those who never use tobacco or nicotine products. The goal is to identify damage that is found at higher levels or remains in the oral cells longer because they might be more important in causing cancer than other types of damage.

DETAILED DESCRIPTION:
DNA damage (adducts) in the oral cells will be measured in people who smoke and vape while they are using their products regularly for two weeks. Then half of the participants will be asked to stop smoking or vaping. Biological samples (saliva, urine, mouth cells, and cheek cells) will be collected at 6 visits to determine how DNA damage changes in the mouth cells of people asked to stop using their products to those who continue to use their product. The DNA damage in these groups will also be compared to those who do not use tobacco or nicotine products at all. It is believed that DNA damage that remains in the cells longer or that is at higher levels than other DNA damage might be more important to cancer formation.

ELIGIBILITY:
Inclusion Criteria:

* 21+ years old
* Good physical and mental health
* Stable physical and mental health
* Either 1) smokes cigarettes daily, 2) vapes daily, 3) does not use any tobacco or nicotine products

Exclusion Criteria:

* Pregnant or nursing
* High blood pressure
* Unstable health condition(s)
* History of cancer or liver disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Oral DNA damage (adduct) levels | DNA damage will be assessed at baseline and Days 3, 6, 12, and 21 after stopping use or continuing use
  The levels and types of DNA damage (adducts) will be measured in the oral cells of all participants. DNA adducts will be reported as fmol/umol dG or as # adducts / 10^8 nucleotides.
  DNA adduct levels will be compared between those who continue to use their products, those who stop using their products, and those who never use tobacco or nicotine products.
  The goal is to identify DNA damage that is found at higher levels or remains in the oral cells longer because they might be more important in causing cancer than other types of DNA damage.
Urinary smoking markers | Urine levels will be measured at baseline and Days 3, 6, 12, and 21 after stopping use or continuing use.
  Total nicotine equivalents (TNE), cyanoethyl mercapturic acid (CEMA), and NNAL will be measured in the urine of participants to confirm if they smoked during the study. The concentration of these compounds will be reported at pmol/mL urine

SECONDARY OUTCOMES:
Urinary vape markers | Vaping markers will be measured in the urine at baseline and Days 3, 6, 12 and 21 after stopping or continuing use.
  Propylene glycol and glycerol will be measured in the urine of participants to confirm if they vaped during the study. The concentration of these compounds will be reported as pmol/mL urine.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hecht, Principal Investigator — University of Minnesota